CLINICAL TRIAL: NCT03384329
Title: Efficacy and Safety of Resveratrol in the Treatment of Depression: Double-blind Randomized Placebo-controlled Parallel-group Study.
Brief Title: Efficacy of Resveratrol in Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Russian Academy of Medical Sciences (Other)
Collaborators: Russian Science Foundation (Other)
Responsible Party: Principal Investigator, Lyubomir I Aftanas, MD, PhD, DrSci., Prof., Director of the Institute of Physiology and Basic Medicine, Principal Investigator, Russian Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RESV-depression
Record Dates: First submitted 2017-12-11; First posted 2017-12-27 (Actual); Results first posted 2020-11-17 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Resveratrol Pill (Experimental)
  Interventions: Drug: Resveratrol Pill
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Resveratrol Pill — Resveratrol 500 mg
  Arms: Resveratrol Pill
Drug: Placebos — Placebo Pills
  Arms: Placebo

SUMMARY:
Patients with depression (target number - 60) receive resveratrol 500 mg or placebo (1:1) each morning daily for 1 month with primary outcome measures of the score change on depression rating scale HDRS-17 and change in SIRT1 activity in the blood measured 4 times over the study period (before, in the middle, after the intervention, and in 2 week follow up).

ELIGIBILITY:
Inclusion Criteria (selectively):

* MDD recurrent or with single episode with melancholic features or dysthymia (DSM-5);
* current depression.

Exclusion Criteria (selectively):

* serious or unstable disease;
* antidepressants intake.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-04 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-09-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Lyubomir I. Aftanas, Novosibirsk, Russia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eight enrolled patients dropped out during the 5-day run-in inpatient-study period
Period: Overall Study
Arm/Group | Resveratrol Pill | Placebo
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Resveratrol Pill | Placebo | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (8.8) | 38.1 (10.8) | 37.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 5 | 5 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 11 | 11 | 22
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 24.3 (4.1) | 22.4 (3.7) | 23.3 (4.0)
Major depressive disorder (MDD) type [Count of Participants; unit: Participants] — recurrent / single / persistent MDD, according to the DSM-5 classification
  Participants
    recurrent | 1 | 6 | 7
    single | 4 | 2 | 6
    persistent | 6 | 3 | 9
Winter season [Number; unit: participants] — Number of participants enrolled/treated in the dark half of the year
  participants | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Total HDRS-17 Score From Baseline to Week 4
Description: Hamilton Depression Rating Scale 17 items, total score range 0-53 (53 - worse)
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resveratrol Pill | Placebo
Number analyzed (Participants) | 11 | 11
score on a scale | -7.2 (5.3) | -9.9 (7.0)

2. Primary Outcome: Change in SIRT1 Activity From Baseline to Week 4
Description: SIRT1 is enzyme sirtuin-1 which activity is measured in the blood
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Resveratrol Pill | Placebo
Number analyzed (Participants) | 11 | 11
units | -0.59 (1.14) | -0.02 (1.58)

3. Secondary Outcome: Change in Total BDI-II Score From Baseline to Week 4
Description: Beck Depression Inventory 21 items, total score range 0-63 (63 - worse)
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resveratrol Pill | Placebo
Number analyzed (Participants) | 11 | 11
score on a scale | -9.3 (11.5) | -9.7 (10.5)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: UKU Side-Effect Rating Scale was used in all 4 visits to collect adverse event information
Arm/Group | Resveratrol Pill | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT03384329/Prot_SAP_000.pdf